CLINICAL TRIAL: NCT03352388
Title: Tailored Food Solutions for Improving Nutrition and Well-being in Older People. Effects on Nutritional and Functional Status and Quality of Life in Older People at Home Care
Brief Title: Effects of Dairy- and Berry-based Snacks on Nutritional and Functional Status and Quality of Life in Older People
Acronym: MAVIRE1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Finland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MAVIRE 247124; 4249/31/2014 (Other Grant/Funding Number: Tekes)
Record Dates: First submitted 2017-11-20; First posted 2017-11-24 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Nutrition Disorders in Old Age
Keywords: Older people; Nutrition; Snack; Dairy; Protein; Berries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Snack (Experimental): Dairy- and berry-based snacks
  Interventions: Dietary Supplement: Dairy- and berry-based snacks
- Reference (No Intervention): No snacks

INTERVENTIONS:
Dietary Supplement: Dairy- and berry-based snacks — High-protein dairy-based products and energy-enriched berry products for three months
  Arms: Snack

SUMMARY:
Malnutrition or its risk is common among older people, especially among those receiving home care services. It impairs the quality of life of the older people and results in significant costs to society. To maintain adequate nutrition, increased meal frequency is important. In addition to main meals, regular consumption of tasty, convenient, nutrient- and energy-dense snacks is recommended. The purpose of this study is to investigate the effects of dairy- and berry-based snack consumption on nutritional and functional status and quality of life among vulnerable older people at home care.

ELIGIBILITY:
Inclusion Criteria:

* Home care clients of the City of Kuopio

Exclusion Criteria:

* Advanced dementia

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 85 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Nutritional status | Baseline and 3 months
  Nutritional status is assessed by the Mini Nutritional Assessment (MNA) test which is a validated and standardized tool for detecting malnutrition and its risk in older people. Scores 24.0 - 30.0 indicate normal nutritional status, scores 17.0 - 23.5 risk of malnutrition and scores < 17.0 malnutrition. Change in the MNA score is determined.
Albumin | Baseline and 3 months
  Change in plasma albumin concentration
Prealbumin | Baseline and 3 months
  Change in plasma prealbumin concentration
Hand grip strength | Baseline and 3 months
  Change in grip strength of both hands

SECONDARY OUTCOMES:
Body mass index (BMI) | Baseline and 3 months
  Change in BMI
Mid-arm muscular area (MMA) | Baseline and 3 months
  Change in MMA
Hemoglobin | Baseline and 3 months
  Change in blood hemoglobin concentration
C-reactive protein (CRP) | Baseline and 3 months
  Change in plasma high-sensitivity CRP concentration
Activity and sleep assessed by ActiGraph monitoring | Baseline and 3 months
  Changes in several parameters describing physical activity and quality of sleep
Health-related quality of life | Baseline and 3 months
  Health-related quality of life is assessed by the 15D instrument. It is a generic, standardized instrument consisting of 15 dimensions: moving, vision, hearing, breathing, sleeping, eating, speech, elimination, usual activities, mental functioning, discomfort/symptoms, depression, distress, vitality, and sexual activity. Each dimension is divided into five levels by which more or less an attribute is distinguished. In this study 15D is used as single index score measure. The single index score (15D score) is calculated from the health state descriptive system through the use of an additive three-stage valuation model based on the multiattribute utility theory. The preference weights for the 15 dimensions, and their levels have been elicited from representative population samples. The 15D score is on a 0-1 scale, where 1 stands for "full health" and 0 being dead. Change in the 15D score is determined, and a change of ±.03 is clinically important.

CONTACTS AND LOCATIONS:
Overall Officials: Riitta Törrönen, PhD, Principal Investigator — Senior Researcher; Irma Nykänen, PhD, Principal Investigator — Senior Researcher; Ursula Schwab, PhD, Principal Investigator — Professor; Mika Tarvainen, PhD, Principal Investigator — Senior Researcher
Locations (1):
- University of Eastern Finland, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nykanen I, Torronen R, Schwab U. Dairy-Based and Energy-Enriched Berry-Based Snacks Improve or Maintain Nutritional and Functional Status in Older People in Home Care. J Nutr Health Aging. 2018;22(10):1205-1210. doi: 10.1007/s12603-018-1076-7. PMID 30498827